CLINICAL TRIAL: NCT02246088
Title: Effect of Neuroscience Education on Subjects With Chronic Knee Pain Related to Osteoarthritis : a Randomized Controlled Trial
Brief Title: Neuroscience Education on Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Valencia (Other)
Collaborators: Hospital de la Ribera (Other)
Responsible Party: Principal Investigator, Enrique Lluch Girbés, Physiotherapist, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EDUART13
Record Dates: First submitted 2014-09-15; First posted 2014-09-22 (Estimated); Last update posted 2014-09-22 (Estimated); Status verified 2014-09

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis, Central Nervous System Sensitization
MeSH Terms: conditions — Osteoarthritis | interventions — NADH dehydrogenase subunit 4

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MT + NE (Experimental): A manual therapy (MT) intervention combined with neuroscience education (NE)
  Interventions: Procedure: MT + NE
- MT + E (Active Comparator): Manual therapy (MT) intervention plus an educational program based on a traditional patho-anatomical or biomedical model (E)
  Interventions: Procedure: MT + E

INTERVENTIONS:
Procedure: MT + NE — Manual therapy will be applied using mobilization with movement (MWM) techniques. MWM will consist of a sustained manual glide of the tibia (either medial, lateral, anterior, posterior, or rotation) during active knee flexion and extension, depending on which are the limited/painful movements for each patient.
  The content and pictures of the neuroscience education (NE) will be based on the text "Explicando el dolor" (Spanish version of "Explain Pain").
  Arms: MT + NE
Procedure: MT + E — Program of education based on the traditional biomedical model (i.e. through visualization of several videos related to anatomy, biomechanics and surgical procedure of the knee), plus the same manual treatment as per the MT+NE group
  Arms: MT + E

SUMMARY:
Osteoarthritis (OA) is a frequent chronic musculoskeletal pathology that usually causes great disability and significant healthcare costs. Substantial scientific evidence indicates a role for central sensitization in OA pain. Reconceptualization of pain through Neuroscience Education (NE) is an intervention that has already been used successfully in some chronic musculoskeletal pain conditions characterized by alteration on CNS pain processing or central sensitization (i.e. chronic low back pain, chronic fatigue syndrome, widespread pain and chronic whiplash associate disorders).There is compelling evidence that NE have a positive effect on pain, disability, catastrophization and physical performance for chronic musculoskeletal pain disorders, yet studies examining the value of NE for OA patients are essentially lacking.

The primary aim of this study is to assess the effect of NE on pain, disability and physical performance in subjects with chronic OA knee pain waiting for replacement surgery. This will be the first time NE will be addressed specifically to OA pain. To investigate the benefits of NE on pain related to knee OA, the effect of a manual therapy intervention combined with NE (MT+NE) will be compared with this same manual intervention plus an educational program based on a traditional patho-anatomical or biomedical model (MT+E). The following secondary aims will be addressed as well:

* Examining the effects of the two interventions on the mechanism of central sensitization in patients with knee OA;
* Examining the effects of the two interventions on pain catastrophizing, illness perceptions and kinesiophobia in patients with knee OA;
* Finally, it is aimed at identifying effect moderators for NE in patients with knee OA.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a frequent chronic musculoskeletal pathology that usually causes great disability and significant healthcare costs. Substantial scientific evidence indicates a role for central sensitization in OA pain. Pathophysiological mechanisms underlying central sensitisation are complex and numerous, but the net effect is an amplification of neural signaling within the CNS than elicits pain hypersensitivity. Central sensitization management is an area of great interest at least in a subgroup of patients with OA pain.

Reconceptualization of pain through Neuroscience Education (NE) is an intervention that has already been used successfully in some chronic musculoskeletal pain conditions characterized by alteration on CNS pain processing or central sensitization (i.e. chronic low back pain, chronic fatigue syndrome, widespread pain and chronic whiplash associate disorders). Moreover, some clinical guides to help clinicians to identify and explain central sensitization through NE, have been recently published. However, this kind of intervention has never been tested specifically for chronic pain related to OA.

Preoperative education centered on a biomedical model of anatomy and pathoanatomy as well as procedural information has limited effect in reducing postoperative pain after total hip arthroplasty and total hip arthroplasty surgeries. Preoperative educational sessions that aim to increase patient knowledge of pain science (i.e. NE) may be more effective in managing postoperative pain. NE is a cognitive-based educational intervention that aims to reduce pain and disability by helping patients gain an increased understanding of the biological processes underpinning their pain state. There is compelling evidence that NE have a positive effect on pain, disability, catastrophization and physical performance for chronic musculoskeletal pain disorders, yet studies examining the value of NE for OA patients are essentially lacking.

Joint mobilization has been shown to be a useful modality to reduce pain related to osteoarthritis. Regarding the knee joint, two recent systematic reviews demonstrated the usefulness of manual therapy and exercise for the management of knee OA. Moreover, Deyle et al reported a preliminary clinical prediction rule which may help to identify the minority of knee OA patients who are unlikely to respond to this management approach.

The primary aim of this study is therefore to assess the effect of NE on pain, disability and physical performance in subjects with chronic OA knee pain waiting for replacement surgery. This will be the first time NE will be addressed specifically to OA pain. To investigate the benefits of NE on pain related to knee OA, the effect of a manual therapy intervention combined with NE (MT+NE) will be compared with this same manual intervention plus an educational program based on a traditional patho-anatomical or biomedical model (MT+E). The following secondary aims will be addressed as well:

* Examining the effects of the two interventions on the mechanism of central sensitization in patients with knee OA;
* Examining the effects of the two interventions on pain catastrophizing, illness perceptions and kinesiophobia in patients with knee OA;
* Finally, it is aimed at identifying effect moderators for NE in patients with knee OA.

ELIGIBILITY:
Inclusion Criteria:

1. An established diagnosis of knee OA according to American College of Rheumatology criteria and Kellgreen/Lawrence scale grades.
2. To be in a waiting list and scheduled to undergo primary knee arthroplasty.
3. To have sufficient Spanish language skills to comprehend all explanations and to complete the assessment tools.

Exclusion Criteria:

1. Previous knee joint replacement surgery of the affected joint or any other lower limb surgery within the past 6 months.
2. Stated inability to attend or complete the proposed course of intervention and follow-up schedule.
3. Presence of co-morbidities associated with cognitive impairment.
4. Co-existing inflammatory, metabolic, neurological or severe medical conditions, defined as a diagnosis in the medical record severe enough that the patient cannot participate fully in the study procedures (i.e. cardiovascular disease).
5. Functional illiteracy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2013-12; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Endogenous analgesia through the experimental protocol of conditioned pain modulation | Up to 3 months
  For assessing endogenous analgesia, the method examining the influence of the Diffuse Noxious Inhibitory Control system (or spatial summation) on temporal summation will be applied. Recently, the term conditioned pain modulation has been recommended to describe the psychophysical paradigm of Diffuse Noxious Inhibitory Control system in humans

SECONDARY OUTCOMES:
Pain at rest and in the last 24 hours | Up to 3 months
  Participants will be asked to rate their pain at rest and in the last 24 hours on a horizontal 100-mm visual analogue scale (VAS). The horizontal line anchors will be "no pain" and "worst imaginable pain". The VAS is a valid and reliable instrument compared with other pain rating scales and has been well established in clinical practice and research for measuring pain levels in arthritis populations.
Pressure Pain Thresholds | Up to 3 months
  Local and distant sites will be chosen for pressure pain threshold measurement. Regarding local sites, two points will be measured from the knee, 3 cm medial and lateral to the midpoint of the medial and lateral edge of patella, respectively. Regarding control site, a distant site will be used to assess systematic analgesic effect of NE at 5 cm distal to lateral epicondyle.
Western Ontario and McMaster osteoarthritis index (WOMAC scale) | Up to 3 months
  WOMAC assesses pain, stiffness and physical function and can be completed in less than 5 minutes. It's a widely used, reliable, valid and responsive measure of outcome in people with osteoarthritis of the hip or knee.
Health-related quality of life using the self-reported Spanish version SF-36 questionnaire | Up to 3 months
Tampa Scale of Kinesiophobia (TSK) (Spanish version) | Up to 3 months
Pain Catastrophization Scale (PCS) (Spanish version) | Up to 3 months
Chronic Pain Coping Inventory-42 (Spanish version) | Up to 3 months
Chronic Pain Acceptance Questionnaire (Spanish version) | Up to 3 months
Goniometric assessment of knee flexion and extension range of motion | Up to 3 months
Strength of the hamstrings and quadriceps muscles | Up to 3 months
Timed "Up & Go" (TUG) Test | Up to 3 months
  Participants will be required to rise from a standard arm chair, walk at a safe and comfortable pace to a mark 3 m away and then return to a sitting position in the chair. The outcome of the test will be the time to complete the task. Time will be measured on a stopwatch to the nearest one-hundredth of a second.
Central Sensitization Inventory | Up to 3 months
  Signs and symptoms suggesting central sensitization will be monitorized using the Central Sensitization Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Lluch, PT, Principal Investigator — University of Valencia; Luis Aguilella, PhD, Principal Investigator — Hospital Universitario de la Ribera, Alcira (Valencia)
Locations (1):
- Hospital Universitario de La Ribera, Alzira, Valencia, Spain

REFERENCES:
- [Background] Lluch E, Torres R, Nijs J, Van Oosterwijck J. Evidence for central sensitization in patients with osteoarthritis pain: a systematic literature review. Eur J Pain. 2014 Nov;18(10):1367-75. doi: 10.1002/j.1532-2149.2014.499.x. Epub 2014 Apr 3. PMID 24700605
- [Background] Lluch Girbes E, Meeus M, Baert I, Nijs J. Balancing "hands-on" with "hands-off" physical therapy interventions for the treatment of central sensitization pain in osteoarthritis. Man Ther. 2015 Apr;20(2):349-52. doi: 10.1016/j.math.2014.07.017. Epub 2014 Aug 14. PMID 25169787
- [Background] Lluch Girbes E, Nijs J, Torres-Cueco R, Lopez Cubas C. Pain treatment for patients with osteoarthritis and central sensitization. Phys Ther. 2013 Jun;93(6):842-51. doi: 10.2522/ptj.20120253. Epub 2013 Feb 7. PMID 23392185
- [Background] Staud R. Evidence for shared pain mechanisms in osteoarthritis, low back pain, and fibromyalgia. Curr Rheumatol Rep. 2011 Dec;13(6):513-20. doi: 10.1007/s11926-011-0206-6. PMID 21833699
- [Background] Mease PJ, Hanna S, Frakes EP, Altman RD. Pain mechanisms in osteoarthritis: understanding the role of central pain and current approaches to its treatment. J Rheumatol. 2011 Aug;38(8):1546-51. doi: 10.3899/jrheum.100759. Epub 2011 Jun 1. PMID 21632678
- [Background] Lee YC, Nassikas NJ, Clauw DJ. The role of the central nervous system in the generation and maintenance of chronic pain in rheumatoid arthritis, osteoarthritis and fibromyalgia. Arthritis Res Ther. 2011 Apr 28;13(2):211. doi: 10.1186/ar3306. PMID 21542893
- [Background] Arendt-Nielsen L, Nie H, Laursen MB, Laursen BS, Madeleine P, Simonsen OH, Graven-Nielsen T. Sensitization in patients with painful knee osteoarthritis. Pain. 2010 Jun;149(3):573-581. doi: 10.1016/j.pain.2010.04.003. Epub 2010 Apr 24. PMID 20418016
- [Background] Sofat N, Ejindu V, Kiely P. What makes osteoarthritis painful? The evidence for local and central pain processing. Rheumatology (Oxford). 2011 Dec;50(12):2157-65. doi: 10.1093/rheumatology/ker283. Epub 2011 Sep 27. PMID 21954151
- [Background] Woolf CJ. Central sensitization: implications for the diagnosis and treatment of pain. Pain. 2011 Mar;152(3 Suppl):S2-S15. doi: 10.1016/j.pain.2010.09.030. Epub 2010 Oct 18. PMID 20961685
- [Background] Murphy SL, Lyden AK, Phillips K, Clauw DJ, Williams DA. Subgroups of older adults with osteoarthritis based upon differing comorbid symptom presentations and potential underlying pain mechanisms. Arthritis Res Ther. 2011 Aug 24;13(4):R135. doi: 10.1186/ar3449. PMID 21864381
- [Background] Moseley L. Combined physiotherapy and education is efficacious for chronic low back pain. Aust J Physiother. 2002;48(4):297-302. doi: 10.1016/s0004-9514(14)60169-0. PMID 12443524
- [Background] Moseley L. Unraveling the barriers to reconceptualization of the problem in chronic pain: the actual and perceived ability of patients and health professionals to understand the neurophysiology. J Pain. 2003 May;4(4):184-9. doi: 10.1016/s1526-5900(03)00488-7. PMID 14622702
- [Background] Moseley GL, Nicholas MK, Hodges PW. A randomized controlled trial of intensive neurophysiology education in chronic low back pain. Clin J Pain. 2004 Sep-Oct;20(5):324-30. doi: 10.1097/00002508-200409000-00007. PMID 15322439
- [Background] Ryan CG, Gray HG, Newton M, Granat MH. Pain biology education and exercise classes compared to pain biology education alone for individuals with chronic low back pain: a pilot randomised controlled trial. Man Ther. 2010 Aug;15(4):382-7. doi: 10.1016/j.math.2010.03.003. Epub 2010 Mar 31. PMID 20359937
- [Background] Meeus M, Nijs J, Van Oosterwijck J, Van Alsenoy V, Truijen S. Pain physiology education improves pain beliefs in patients with chronic fatigue syndrome compared with pacing and self-management education: a double-blind randomized controlled trial. Arch Phys Med Rehabil. 2010 Aug;91(8):1153-9. doi: 10.1016/j.apmr.2010.04.020. PMID 20684894
- [Background] Van Oosterwijck J, Nijs J, Meeus M, Truijen S, Craps J, Van den Keybus N, Paul L. Pain neurophysiology education improves cognitions, pain thresholds, and movement performance in people with chronic whiplash: a pilot study. J Rehabil Res Dev. 2011;48(1):43-58. doi: 10.1682/jrrd.2009.12.0206. PMID 21328162
- [Background] Clarke CL, Ryan CG, Martin DJ. Pain neurophysiology education for the management of individuals with chronic low back pain: systematic review and meta-analysis. Man Ther. 2011 Dec;16(6):544-9. doi: 10.1016/j.math.2011.05.003. Epub 2011 Jun 25. PMID 21705261
- [Background] Louw A, Puentedura EL, Mintken P. Use of an abbreviated neuroscience education approach in the treatment of chronic low back pain: a case report. Physiother Theory Pract. 2012 Jan;28(1):50-62. doi: 10.3109/09593985.2011.562602. Epub 2011 Jul 3. PMID 21721995
- [Background] Nijs J, Van Houdenhove B, Oostendorp RA. Recognition of central sensitization in patients with musculoskeletal pain: Application of pain neurophysiology in manual therapy practice. Man Ther. 2010 Apr;15(2):135-41. doi: 10.1016/j.math.2009.12.001. Epub 2009 Dec 24. PMID 20036180
- [Background] Nijs J, Paul van Wilgen C, Van Oosterwijck J, van Ittersum M, Meeus M. How to explain central sensitization to patients with 'unexplained' chronic musculoskeletal pain: practice guidelines. Man Ther. 2011 Oct;16(5):413-8. doi: 10.1016/j.math.2011.04.005. Epub 2011 May 31. PMID 21632273
- [Background] Louw A, Diener I, Butler DS, Puentedura EJ. Preoperative education addressing postoperative pain in total joint arthroplasty: review of content and educational delivery methods. Physiother Theory Pract. 2013 Apr;29(3):175-94. doi: 10.3109/09593985.2012.727527. Epub 2012 Oct 4. PMID 23035767
- [Background] Louw A, Diener I, Butler DS, Puentedura EJ. The effect of neuroscience education on pain, disability, anxiety, and stress in chronic musculoskeletal pain. Arch Phys Med Rehabil. 2011 Dec;92(12):2041-56. doi: 10.1016/j.apmr.2011.07.198. PMID 22133255
- [Background] Moss P, Sluka K, Wright A. The initial effects of knee joint mobilization on osteoarthritic hyperalgesia. Man Ther. 2007 May;12(2):109-18. doi: 10.1016/j.math.2006.02.009. Epub 2006 Jun 13. PMID 16777467
- [Background] Takasaki H, Hall T, Jull G. Immediate and short-term effects of Mulligan's mobilization with movement on knee pain and disability associated with knee osteoarthritis--a prospective case series. Physiother Theory Pract. 2013 Feb;29(2):87-95. doi: 10.3109/09593985.2012.702854. Epub 2012 Jul 30. PMID 22844980
- [Background] French HP, Brennan A, White B, Cusack T. Manual therapy for osteoarthritis of the hip or knee - a systematic review. Man Ther. 2011 Apr;16(2):109-17. doi: 10.1016/j.math.2010.10.011. Epub 2010 Dec 13. PMID 21146444
- [Background] Jansen MJ, Viechtbauer W, Lenssen AF, Hendriks EJ, de Bie RA. Strength training alone, exercise therapy alone, and exercise therapy with passive manual mobilisation each reduce pain and disability in people with knee osteoarthritis: a systematic review. J Physiother. 2011;57(1):11-20. doi: 10.1016/S1836-9553(11)70002-9. PMID 21402325
- [Background] Deyle GD, Gill NW, Allison SC, Hando BR, Rochino DA. Knee OA: which patients are unlikely to benefit from manual PT and exercise? J Fam Pract. 2012 Jan;61(1):E1-8. PMID 22220299
- [Derived] Huysmans E, Baeyens JP, Duenas L, Falla D, Meeus M, Roose E, Nijs J, Lluch Girbes E. Do Sex and Pain Characteristics Influence the Effectiveness of Pain Neuroscience Education in People Scheduled for Total Knee Arthroplasty? Secondary Analysis of a Randomized Controlled Trial. Phys Ther. 2021 Dec 1;101(12):pzab197. doi: 10.1093/ptj/pzab197. PMID 34459493